CLINICAL TRIAL: NCT04835883
Title: Open-label, Single-arm, 24-week Investigator Study to Evaluate the Efficacy and Safety of CS20AT04 (HLA-haplo Matched Allogenic Bone Marrow-Derived Stem Cells) Administered in Patients With Lupus Nephritis or Lupus Cytopenia
Brief Title: Exploring the Efficacy and Safety of CS20AT04 (Allogenic Bone Marrow-Derived Stem Cell) in Systemic Lupus Erythematosus Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanyang University Seoul Hospital (Other)
Collaborators: Corestemchemon, Inc. (Industry); Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Chan-Bum Choi, Principal Investigator, Hanyang University Seoul Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS20AT04-SLE101
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; Allogenic bone marrow-derived mesenchymal stem cell; Lupus Nephritis; Lupus Cytopenia; Cell Therapy; Phase IIa Clinical Trial
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned interventions (Experimental): Subjects enrolled into the CS20AT04 with corticosteroid taper regimen arm will receive two infusions of CS20AT04 (2.0×10^6cell/kg), on 0 day and on 12 weeks post-enrollment.
  Interventions: Biological: CS20AT04 (allogenic bone marrow derived mesenchymal stem cell)

INTERVENTIONS:
Biological: CS20AT04 (allogenic bone marrow derived mesenchymal stem cell) — Two intravenous infusions of CS20AT04 (2.0×10^6cell/kg), on 0 day and on 12 weeks The target population of this study is subjects in South Korea with a diagnosis of either lupus nephritis or lupus cytopenia.

SUMMARY:
This is an open-label, one-arm single-center phase Ⅱa study exploring the efficacy and safety of CS20AT04 (HLA-haplo Matched Allogenic Bone Marrow-Derived Stem Cells) in two subpopulation group of systemic lupus erythematosus patients - lupus nephritis and lupus cytopenia.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic inflammatory disease of unknown cause that can affect virtually every organ. A subset of SLE patients continues to suffer significant morbidity and mortality from active disease, with visceral organ involvement. Therefore, it is urgent to develop a more effective therapy for SLE disorder, especially for treatment-refractory patients.

Bone marrow-derived mesenchymal stem cells are known to be effective in modulating immune cells such as T lymphocytes, B lymphocytes, dendritic cells, and Neutral Killer (NK) cells and treating acute Graft-Versus-Host Disease (GVHD). Also, based on the anti-inflammatory and immunomodulatory properties, bone marrow-derived mesenchymal stem cells have been widely studied as a candidate for the treatment of refractory immune- and inflammation-mediated disease, and have extensive experience of use.

Half-matched allogeneic bone marrow-derived mesenchymal stem cells, the active ingredient of CS20AT04 Injection, not only have the potential to differentiate into various mesenchymal cells but also have various immunomodulatory and anti-inflammatory effects, and thus are expected to induce and maintain remission of lupus nephritis and lupus cytopenia.

This study is designed to investigate the following. Subjects enrolled into the CS20AT04 with corticosteroid taper regimen arm will receive two infusions of CS20AT04(2.0×10^6cell/kg), on 0 day and on 12 weeks post-enrollment. Subjects will return for efficacy and safety assessments on 3 days, 1 week, and every 4 weeks each post-infusion until Week 24. Safety monitoring will be continued at 1 year, 3 years, and 5 years post-infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HLA-haplo-matched bone marrow donor less than 70 years old
2. Patients meeting:

   -at least 4 of the 2012 Systemic Lupus International Collaborating Clinics (SLICC) criteria, including at least 1 clinical criterion and 1 immunology criterion; or

   -at least 4 of the 11 Revised American College of Rheumatology (ACR) Criteria for Classification of Systemic Lupus Erythematosus, according to the 1997 Update of the 1982 ACR
3. Patients having a positive test result for antinuclear antibody (ANA; titer at least 1:80) and/or anti-double stranded DNA antibody (anti-dsDNA Ab) at screening
4. Patients (non-responder or partial responder), defined as :

   -unresponsive to treatment with standard care(such as monthly i.v. pulse cyclophosphamide (CYC) 500-1000 mg/m2, mycophenolate (MMF) ≥ 2 gm/day, azathioprine (AZA) ≥ 200 mg/day, leflunomide (LEF) 20 mg/day, oral CYC, cyclosporine, mizoribine ≥ 150 mg/day, mycophenolic acid ≥ 1.44 g/day, tacrolimus (TAC) ≥ 1.5 mg twice a day alone or in combination for at least 6 months) or

   -with continued daily dosage of ≥15mg of prednisone or its equivalent for maintenance treatment

   5-1. For the lupus cytopenia sub-group only:
   * Patients with refractory cytopenia (at least one of anemia, leukopenia, or thrombocytopenia) in absence of any other identifiable cause, defined as:

   [Red blood cell associated] -Hemolytic anemia (Hgb ≤ 10g/dL) with reticulocytosis, or [White cell associated]

   -Neutrophil count < 1,000/mm3 (in the absence of other known cause such as corticosteroids, drugs, and infection), and/or
   * Lymphocyte count < 1,500/mm3 [Platelet associated]
   * Platelet count < 100,000/mm3 (in the absence of other known cause such as drugs, portal hypertension, and thrombotic thrombocytopenic purpura (TTP))

   5-2. For the lupus nephritis sub-group only: •Patients with clinical disease activity of lupus nephritis, defined by:
   * laboratory tests documented active lupus nephritis three consecutive times: (i) decrease in renal function (serum creatinine > 106 μmol/L) (ii) increase in proteinuria (defined as urine protein/creatinine ratio (UPC) > 1), and (iii) deterioration in microscopic hematuria (defined as > 10 red cells per high power field) in the absence of menstrual hematuria or urinary tract infection at the time of screening or the presence of cellular casts
   * renal biopsy documenting lupus nephritis according to the International Society of Nephrology/Renal Pathology Society classification of active or active/chronic lupus nephritis in renal biopsy class III, class IV-S or IV-G, class V, class III + V, or class IV + V (within 1 year)

   Exclusion Criteria:

1. Patients unable or unwilling to provide written informed consent

2. Patients with any history of cancer, allergy, alcohol or substance abuse, active peptic ulcer disease, heart failure, liver disease, and coagulation disorder

3. Patients who have active severe central nervous system (CNS) lupus

4. Patients who have received biologic investigational agents in the past year

5. Patients undergoing intravenous immunoglobulin or plasma exchange therapy

6. Patients who are pregnant or are lactating

7. Patients with any evidence of a major infection

8. For the lupus nephritis sub-group only: Patients with serum creatinine > 250 μmol/L

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-11-05 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Reduction of corticosteroid dose to ≤ 7.5 mg/day of prednisone or equivalent | 24 weeks
  The primary efficacy objective of this study is to assess the efficacy of CS20AT04, in combination with a 24-week corticosteroid taper regimen, as measured by:
  Reduction of corticosteroid dose to ≤ 7.5 mg/day of prednisone or equivalent at Week 4 , and continued through Week 12
Hematologic improvement without ongoing SLE treatment | 24 weeks
  As Lupus cytopenia sub-group specific endpoint, Hgb increase of ≥ 1.5 g/dL, or Neutrophil count increase of ≥ 100% from pre-treatment level and an absolute increase of 500/mm3 x 10^9/L, or For pre-treatment platelet count > 20 X 10^9/L, a platelet absolute increase of ≥ 30 X 10^9/L For pre-treatment platelet count ≤ 20 X 10^9/L, a platelet absolute increase ≥ 20 X 10^9/L and ≥ 100% increase from pre-treatment level
Renal response improvement | 24 weeks
  As Lupus nephritis (LN) sub-group specific endpoint, a renal response at 24 weeks adjudicated based on the following parameters:
  Urine Protein to Creatinine Ratio (UPCR) of ≤0.5mg/mg, and Estimated Glomerular Filtration Rate (eGFR)≥60mL/min/1.73m2 or no confirmed decrease from baseline in eGFR of > 20%, and Did not receive any rescue medication for LN, and Did not receive over than 7.5mg prednisone for ≥7 consecutive days in total during week 12 through 24, just prior to the renal response assessment

SECONDARY OUTCOMES:
Proportion of subjects who achieve a prednisone dose of ≤ 7.5mg/day or equivalent | 12 weeks, 24 weeks
  Proportion of subjects who achieve a prednisone dose of ≤ 7.5mg/day or equivalent by Week 12 and maintain this dose ≤ 7.5mg/day prednisone or equivalent from Week 12 to 24
Proportion of subjects achieving Low Level Disease Activity State | 24 weeks
  Proportion of subjects achieving Low Level Disease Activity State (LLDAS) at Week 24
Proportion of subjects with ≥ 4 point reduction from baseline in Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K) score | 24 weeks
  Proportion of subjects with ≥ 4 point reduction from baseline in SLEDAI-2K score at 24 weeks
Proportion of subjects with baseline Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K) ≥ 4 having SLE responder index 4 (SRI5) | 24 weeks
  Proportion of subjects with baseline SLEDAI-2K ≥ 4 having SLE responder index 5 (SRI5) response at 24 weeks, defined by (i) a ≥ 4 point reduction from baseline in SLEDAI-2K score, (ii) no worsening (increase of < 0.30 points from baseline) in Physician's Global Assessment (PGA), and (iii) no new British Isles Lupus Assessment Group of SLE Clinics (BILAG) A organ domain score or 2 new BILAG B organ domain scores compared with baseline at the time of assessment (i.e. at 24 weeks)
Proportion of subjects with baseline Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K) ≥ 5 having SLE responder index 5 (SRI5) | 24 weeks
  Proportion of subjects with baseline SLEDAI-2K ≥ 5 having SLE responder index 5 (SRI5) response at 24 weeks, defined by (i) a ≥ 5 point reduction from baseline in SLEDAI-2K score, (ii) no worsening (increase of < 0.30 points from baseline) in Physician's Global Assessment (PGA), and (iii) no new British Isles Lupus Assessment Group of SLE Clinics (BILAG) A organ domain score or 2 new BILAG B organ domain scores compared with baseline at the time of assessment (i.e. at 24 weeks)
Proportion of subjects with baseline Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K) ≥ 6 having SLE responder index 6 (SRI6) | 24 weeks
  Proportion of subjects with baseline SLEDAI-2K ≥ 6 having SRI6 response at 24 weeks, defined by (i) a ≥ 6 point reduction from baseline in SLEDAI-2K score, (ii) no worsening (increase of < 0.30 points from baseline) in Physician's Global Assessment (PGA), and (iii) no new British Isles Lupus Assessment Group of SLE Clinics (BILAG) A organ domain score or 2 new BILAG B organ domain scores compared with baseline at the time of assessment (i.e. at 24weeks)
Time to first severe modified SLE Flare Index (SFI) flare | 24 weeks
  Time to first severe modified SLE Flare Index (SFI) flare over 24 weeks
Change from baseline of hematologic parameters | 3 days, 1 week, 4 weeks, 12 weeks , and 24 weeks
  For the lupus cytopenia sub-group only: Change from baseline of hematologic parameters (white blood cell counts, platelet counts, and hemoglobin) at 3 days, 1 week, 4 weeks, 12 weeks, and 24 weeks
Time to first hematologic flare | 24 weeks
  For the lupus cytopenia sub-group only: Time to first hematologic flare over 24 weeks
Change in baseline of renal function parameters | 24 weeks
  For the lupus nephritis sub-group only:
  Time to event for each of the individual components of treatment failure (death, ESRD, sustained doubling of serum creatinine, renal flare, extrarenal flare, or rescue therapy)
Time to event for each of the individual components of treatment failure | 24 weeks
  For the lupus nephritis sub-group only:
  Time to event for each of the individual components of treatment failure (death, End-Stage Renal Disease (ESRD), sustained doubling of serum creatinine, renal flare, extrarenal flare, or rescue therapy)
Time to complete remission | 24 weeks
  For the lupus nephritis sub-group only:
  Time to complete remission over 24 weeks, as defined by return to normal values of serum creatinine (< 106 μmol/L), proteinuria (< 0.3 g/24 h), and urine sediment.
Time to first renal flare | 24 weeks
  For the lupus nephritis sub-group only: Time to first renal flare over 24 weeks

OTHER OUTCOMES:
Change in SLE parameters compare to baseline | 3 days, 1 week, 4 weeks, 12 weeks, and 24 weeks
  Change in the following SLE parameters compared to baseline at 3 days, 1 week, 4 weeks, 12 weeks, and 24 weeks:
  * Total Systemic Lupus Erythematosus Disease Activity Index- 2000 (SLEDAI-2K) score
  * Systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index (SLICC/ACR-DI) score
  * British Isles Lupus Assessment Group (BILAG) scale (at 4 weeks, 12 weeks, and 24 weeks)
Change from baseline of Treg CD4+CD25+Foxp3+) and Th17 (CD3+CD8-IL-17A+) cell counts | 3 days, 1 week, 4 weeks, 12 weeks, 24 weeks and 0.5 years, 1 year, 1.5 years, 2 years, 3 years
  Change from baseline of Treg (CD4+CD25+Foxp3+) and Th17 (CD3+CD8-IL-17A+) cell counts at 3 days, 1 week, 4 weeks, 12 weeks, 24 weeks and 0.5 years, 1 year, 1.5 years, 2 years, 3 years after the first injection, as measured by flow cytometry (FACS) analysis
  * CD=Cluster of Differentiation, Foxp=forkhead box P, IL=Interleukin

CONTACTS AND LOCATIONS:
Overall Officials: Chan-Bum Choi, M.D.,Ph.D., Principal Investigator — Department of Rhumatology in Hanyang University Medical Center
Locations (1):
- Hanyang University Medical Center, Seoul, South Korea